CLINICAL TRIAL: NCT05379660
Title: Effects of Transcutaneous Electrical Acupoint Stimulation on Postoperative Recovery of Intestinal Function in Children Undergoing Laparoscopic Appendectomy
Brief Title: Effects of TEAS on Postoperative Recovery of Intestinal Function in Children Undergoing Laparoscopic Appendectomy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Xian Children's Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: 2021-015-01
Record Dates: First submitted 2022-05-04; First posted 2022-05-18 (Actual); Last update posted 2022-05-18 (Actual); Status verified 2022-05

CONDITIONS: Transcutaneous Electrical Acupoint Stimulation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- T1 treatment group (Experimental): TEAS initiates at 30 minutes before induction and lasts for 30 minutes
  Interventions: Device: transcutaneous electrical acupoint stimulation
- T2 treatment group (Experimental): TEAS initiates immediately after skin incision and lasts for 30 minutes
  Interventions: Device: transcutaneous electrical acupoint stimulation
- T3 treatment group (Experimental): TEAS initiates immediately after extubating and lasts for 30 minutes
  Interventions: Device: transcutaneous electrical acupoint stimulation
- control group (No Intervention): Electrodes are placed on the same acupoints, but no current is given

INTERVENTIONS:
Device: transcutaneous electrical acupoint stimulation — Basing on the theory of traditional Chinese medicine, bilateral Zusanli (ST 36), Shangjuxu (ST 37) and Sanyinjiao (SP 6) are elected as the acupuncture points,the electrode pads with wire are attached to the corresponding acupoints, which are connected with Hwato electric acupuncture treatment instrument,TEAS stimulation uses a dense-dispersed wave with frequencies of 2 and 100 Hz alternating every 3 s, and the intensity 5 ~ 12mA,on the first and second days after surgery, the doctor who is responsible for acupuncture will arrive at the ward in the morning and afternoon to administer TEAS stimulation at the same acupoints for 30 min in the TEAS groups
  Arms: T1 treatment group; T2 treatment group; T3 treatment group

SUMMARY:
With the development of surgical techniques, laparoscopic appendectomy has become a standard therapeutic procedure for acute appendicitis in many hospitals in recent years, which is considered as an effective and safe treatment option in children. Even so, patients still experience gastrointestinal dysfunction after surgery, which is one of the most common complications in patients who have undergone major abdominal surgery. The application of laparoscopy reduces trauma in some degree, however, postoperative nausea and vomiting (PONV), abdominal distension, fart, and delayed bowel movement caused by postoperative gastrointestinal dysfunction(PGD), severely disturb patients and seriously affect the quality of patients' postoperative recovery. Previous studies have shown that the incidence of PGD can be as high as 10%-30%. For PGD, the main treatment options include the use of gastric dynamics promoting drug, non-steroidal anti-inflammatory drug, gastrointestinal (GI) decompression, nutritional support, and so forth. However, the effect of these treatments is limited, and there are varying degrees of adverse reactions, which indirectly leads to the low satisfaction of patients. Acupuncture is a form of traditional Chinese medicine and has unique advantages in the treatment of PGD, which have gradually obtained more acceptance from physicians as an alternative therapy. While transcutaneous electrical acupoint stimulation (TEAS) is one of the acupuncture-related technologies and can allow for accurate control of stimulation parameters. For this reason, it is helpful for quantitative research and widely practiced in China. Many studies have shown that TEAS combining with anesthetics can significantly enhance the analgesic effect and reduce the dosage of anesthetics, and can offer certain beneficial effects, such as alleviating preoperative anxiety and reducing postoperative pain and PONV by lessening need for anesthetic usage. It also has been found to help protect the brain, heart and other tissues, with positive benefits for gastrointestinal function by regulating vasoactive intestinal peptide levels. In practice, however, the current TEAS study focused on adults，with relatively little research on their use in children. Because of that, we applied TEAS for use in our study to observe the effect of TEAS in children's laparoscopic surgery and explore its possible mechanism.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists grade I&II,16kg/m2 ≤BMI≤30kg/m2, undergoing laparoscopic appendectomy

Exclusion Criteria:

* previous history of gastrointestinal surgery or abnormal anesthesia recovery, allergy, broken and infection skin at and around the related points, long-term use of analgesic and sedative drugs, presence of severe systemic disease,and the patients drop out or are unable to complete a full follow-up for any reason

Ages: 4 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 200 (Estimated)
Dates: Start 2022-06-30 (Estimated); Primary Completion 2022-12-30 (Estimated); Study Completion 2023-04-30 (Estimated)

PRIMARY OUTCOMES:
the time to first bowel sound | until the time point at which the regular bowel sounds are first heard after surgery up to 1 day
  It was heard by the same researcher , and defined as the first time point at which the regular bowel sounds (more than two sounds every minute) are first heard after surgery.

SECONDARY OUTCOMES:
the time to first passage of flatus | an average of 24 hours,from the end of surgery to the time of the patient's first passage of flatus
  This information was obtained with the help of nurse staff and caregivers through questionnaires which were filled out once daily.
the time to first passage of defecation | an average of 24 hours,from the end of surgery to the the time of the patient's first passage of defecation,
  This information was obtained with the help of nurse staff and caregivers through questionnaires which were filled out once daily.
the first time to normal diet intake | within 48 hours after surgery,from the end of surgery to the time when the patient was given normal diet
  It was defined as the time at which the patient was given normal diet after defecation without nausea or vomiting
the first time to mobilization | within 48 hours after surgery,from the end of surgery to the time when the patient is first able to leave bed
  It was defined as the time at which the patient is first able to leave bed
gastroenterological hormones | three time points: before induction of anesthesia, the end of the surgery and the first day after the operation
  To observe changes in serum levels of gastroenterological hormones ,including serotonin (5-HT), vasoactive intestinal peptide (VIP) and Substance P (SP),venous blood(4ml) will be collected from patients
inflammatory factors | three time points: before induction of anesthesia, the end of the surgery and the first day after the operation
  To observe changes in serum levels of inflammatory factors,which contain tumor necrosis factor (TNF)-α and interleukin-10 (IL-10),venous blood(4ml) will be collected from patients

CONTACTS AND LOCATIONS:
Overall Officials: Fang Li Yang, Study Director — Xi 'an children's hospital